CLINICAL TRIAL: NCT03301610
Title: The Impact of Mobile Education Delivery on Postoperative Pain Outcomes
Brief Title: Mobile Educations Effect on Pain Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: George Washington University (Other)
Responsible Party: Principal Investigator, Amber M. Stitz, Clinical Nurse Specialist, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-004771
Record Dates: First submitted 2017-09-13; First posted 2017-10-04 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Total Joint Arthroplasty; Pain, Postoperative
Keywords: Pain Education; Information Delivery; Mobile Application
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This prospective study has been designed as quasi-experimental study. This study seeks to explore both a treatment and control group in efforts to compare outcomes which are dependent on the type of intervention. Study participants will be assigned into one of two study arms, intervention or control, based on random assignment determined by the location they are bedded in hospital. One of two patient care units will offer standard education, the other unit will offer the mobile, iPad based education. The patient care unit to offer the mobile, iPad based education will be selected at random.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Education Delivery (Experimental): The participants in the study arm will receive comprehensive pain management education delivered using mobile iPads at the point of care. The mobile based education modules will be inclusive of the use of the pain rating scale and assessment of pain; communication with healthcare providers; daily expectations for pain and pain management; pharmacologic and non-pharmacologic treatment options; medication side effects and safety; and discharge instructions including safe handling of opioids, disposal, tapering, and when to call the provider. It will also include an interactive pain and discomfort menu, knowledge based questions, and medication tracking log.
  Interventions: Other: Mobile Education Delivery
- Standard verbal and written education (Placebo Comparator): The control group will receive the current standard of care which consists of verbal instruction and pain management educational pamphlets. At a minimum, the patients will receive two educational pamphlets titled Your Pain and Discomfort Management Menu and Communicating About Your Pain. Verbal instruction is nurse dependent. At a minimum the nurse will provide the two pamphlets to the patient and follow-up with the patient to address any questions.
  Interventions: Other: Standard Verbal and Written Education

INTERVENTIONS:
Other: Mobile Education Delivery — Patients will be provided with an iPad on admission to the post-surgical unit and will remain with the patient until discharge. The patient, independently or with the nurse, may use the program at any point during the inpatient care experience. The RN will use the iPad to engage patients in their pain management.
  Arms: Mobile Education Delivery
Other: Standard Verbal and Written Education — Patients will be provided with two pamphlets on pain management on admission to the post-surgical unit. Nurses will follow-up with verbal instruction based on patient need. This will continue through hospital stay. Additional printed education materials are available through the department of patient education and verbal instruction may be tailored based on nursing assessment and patient need.
  Arms: Standard verbal and written education

SUMMARY:
The purpose of this study is to explore the clinical impact of pain management education using a mobile web-based education delivery system compared to standard education delivery. This study seeks to understand the difference between two different education delivery methodologies and the effect on the postoperative pain experience, including participation in treatment plan, knowledge, pain outcomes, and opioid requirements in patients undergoing major hip (THA) and knee (TKA) arthroplasty. It is hypothesized that a real-time, interactive, mobile education system will demonstrate improved pain associated outcomes and higher patient participation when compared to the current standard education delivery method.

ELIGIBILITY:
Inclusion:

* Adult patients
* over the age of 18 years
* undergoing surgical intervention and inpatient care for one of the following procedures:
* total hip arthroplasty (THA) (primary, bilateral, and revision)
* total knee arthroplasty (TKA) (primary, bilateral, unicompartmental, and revision)
* Fluent in the English language

Exclusion:

* Undergoing more complex hip and knee procedures such as:
* implant resections with or without spacer placement
* liner exchange
* THA or unipolar hip arthroplasty related to repair of hip fracture.
* Preexisting physical or cognitive limitations that would hinder their ability to use the mobile application

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Difference in self-reported pain scores | Post-intervention, at the time of discharge from the hospital (between 1 and 5 days post-surgery)
  Scores are measured using a 10 point (Lickert) pain rating scale. The scale ranges from 0 to 10 with the lower score indicating less pain and the higher score indicating greater pain.

SECONDARY OUTCOMES:
Change in pain management knowledge | Pre-intervention (between 1 and 5 days before surgical procedure) and post-intervention, at the time of discharge from the hospital (between 1 and 5 days post-surgery)
  Scores are measured using a modified Patient Pain Questionnaire; 9 knowledge based questions use a ten-point (0-10) ordinal scale to assess patients' agreement or disagreement with specific statements. All items have been formatted so that zero indicates the most positive outcome and a ten indicates the most negative outcome.
Difference in self-reported participation in pain management | Post-intervention, at the time of discharge from the hospital (between 1 and 5 days post-surgery)
  Scores are measured using a 10 point Lickert scale measuring patients perception of participation in pain management/treatment decisions. The scale ranges from 0 to 10 with the lower score indicating less perceived participation and the higher score indicating greater perceived participation.
Difference in post-operative opioid requirements | Post-intervention, at the time of discharge from the hospital (between 1 and 5 days post-surgery)
  Total opioid requirements, converted to morphine milligram equivalents
Difference in usefulness of education | Post-intervention, at the time of discharge from the hospital (between 1 and 5 days post-surgery)
  Scores are measured using a 10 point Lickert rating scale. The scale ranges from 0 to 10 with the lower score indicating lower perceived usefulness and the higher score indicating greater perceived usefulness.
Difference in use of non-pharmacologic pain modalities | Post-intervention, at the time of discharge from the hospital (between 1 and 5 days post-surgery)
  Results are tabulated for a descriptive selection list for patients to report what interventions were used.

CONTACTS AND LOCATIONS:
Overall Officials: Amber M Stitz, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT03301610/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT03301610/ICF_001.pdf